CLINICAL TRIAL: NCT02366832
Title: Percutaneous Image Guided Cryoablation for the Treatment of Refractory Phantom Limb Pain
Brief Title: Cryoablation for Phantom Limb Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, John Prologo, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00078008
Record Dates: First submitted 2015-02-09; First posted 2015-02-19 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Phantom Limb Syndrome
MeSH Terms: conditions — Phantom Limb | interventions — Cryosurgery; Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cryoablation (Experimental): Amputee subjects experiencing phantom limb syndrome (PLS) will receive cryoablation
  Interventions: Procedure: Cryoablation; Device: 17g Galil Medical Ice Sphere cryoablation needle

INTERVENTIONS:
Procedure: Cryoablation — Subjects who respond to lidocaine nerve block will undergo CT guided cryoablation of the affected nerve stump with a 17g Galil Medical Ice Sphere cryoablation needle.
  Other Names: Cryotherapy; Cryosurgery
Device: 17g Galil Medical Ice Sphere cryoablation needle — Under CT guidance, the corresponding nerve will be targeted with a 17g probe. Two freeze-thaw cycles will be undertaken. The probe will be removed and a final scan obtained.

SUMMARY:
The purpose of this study is to determine if treatment with percutaneous cryoablation yields significant differences in the evaluative criteria of Phantom Limb Syndrome (PLS).

DETAILED DESCRIPTION:
This study aims to treat Phantom Limb Syndrome (PLS) with cryoablation of the remaining nerve stumps. The rationale is that because the pain in PLS follows the known distribution of nerves, and because the amputated nerves are known to undergo changes after the surgery that may lead to excessive "firing," that interruption of the nerve impulses will reduce patient pain.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are status post (s/p) amputation of an upper or lower limb. That is, the amputation is not congenital.
* Refractory pain symptoms, following tissue healing(postoperatively, or post injury) are related to amputation as determined by referring physician and investigator, to include: stump pain, phantom pain, unpleasant phantom sensations, and/or undesirable and/or life-limiting kinesthetic sensations. The character, frequency, location, description, and exacerbation or relieving elements will be recorded.

Patients will be questioned as to the location of their sensation, be it pain, movement, burning, tingling, or other. The location of their pain will be correlated with the corresponding proximal nerve stump.

* Positive anesthetic/steroid block, as performed under CT guidance in an analogous fashion to the cryoablation procedure.
* Absence of infection
* Absence of coagulopathy
* Ability and willingness of patient to provide written informed consent

Exclusion Criteria:

* Active infection
* Underlying congenital segmentation or other spinal anomalies that result in differential nerve root pressures
* Significant spinal stenosis interpreted as "severe" on any cross sectional imaging study
* Pregnant or planning to become pregnant
* Immunosuppression
* History or laboratory results indicative of any significant cardiac, endocrine, hematologic, hepatic, immunologic, infectious, metabolic, urologic, pulmonary, gastrointestinal, dermatologic, psychiatric, renal, neoplastic, or other disorder that in the opinion of the Principal Investigator would preclude the safe performance of cryoablation.
* Uncorrectable coagulopathies
* Concurrent participation in another investigational trial involving systemic administration of agents or within the previous 30 days.
* Have undergone a previous surgical intervention - post amputation - that may have altered the target nerve.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-12-16 (Actual); Study Completion 2016-12-16 (Actual)

PRIMARY OUTCOMES:
Feasibility of cryoablation, defined by number of participants, in which cryoablation was performed successfully | Post-Cryoablation
  Feasibility, defined by number of participants, in which cryoablation was performed successfully
Safety of cryoablation procedure, measured by the number of subjects that had cryoablation procedure events (CPEs). | 56 days
  Safety is measured by the number of subjects that had cryoablation procedure events (CPEs). CPEs are device- or procedure-related serious adverse events (SAE) or adverse events (AE) categorized as clinical signs or symptoms of infection (fever), hemorrhage (pain, imaging changes), nerve pain worsening, or toxicity of any kind (confusion, seizure).

SECONDARY OUTCOMES:
Change in pain scores on visual analogue scale (VAS ) | Baseline, day 56
  Change in pain score will be calculated by subtracting the day 56 pain score from the baseline pain score.The pain scores are on a continuous visual analogue scale of 0 to 100 mm. 0 mm = no pain and 100 mm = worst possible pain. The VAS is scored simply by measuring the distance, in mm, from the patient's mark to one of the ends of the line.
Change in quality of life, measured using Roland-Morris Disability Questionnaire (RDQ) | Baseline, day 56
  Quality of life will be measured using Roland-Morris Disability Questionnaire (RDQ); it is a validated measure of physical disability due to low back pain.The best score is 0 (no disability) and worst is 24 (maximum disability).

CONTACTS AND LOCATIONS:
Overall Officials: John D Prologo, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: YouTube Video — https://youtu.be/ORQKe7tTyFo